CLINICAL TRIAL: NCT03088384
Title: The Effect of Therapeutic Ketamine Infusions on the Symptoms of Post-Traumatic Stress Disorder in Combat Veterans
Brief Title: Ketamine Infusion Therapy for PTSD in Combat Veterans
Status: Completed | Type: Observational
Sponsor: Klarisana Physician Services PLLC (Industry)
Responsible Party: Sponsor
Other Study IDs: KRP001
Record Dates: First submitted 2017-02-26; First posted 2017-03-23 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post Traumatic Stress Disorder; PTSD; Combat Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Combat Veterans: Eligible participants must be military veterans who have served in a combat zone as evidenced by documentation on the subject's DD214 (or equivalent if he/she served in a foreign military). Participants must have a diagnosis of post traumatic stress disorder that was as a result of their military combat experience.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Psychological survey instruments administered before and after a series of six low-dose infusions of ketamine.

SUMMARY:
Klarisana is conducting an observational study in San Antonio, Texas to see if there are tangible improvements in the symptoms of post traumatic stress disorder (PTSD) in combat veterans after receiving a series of six low-dose outpatient infusions of ketamine.

DETAILED DESCRIPTION:
The prolonged conflicts in Iraq and Afghanistan have created a very large population of veterans who suffer from severe post traumatic stress disorder (PTSD). This has, in part, contributed to a rate of suicide that many clinicians and concerned citizens find alarming. In the last two decades, there has been some promising evidence coming to light showing that the medication ketamine can potentially suppress and/or alleviate some of the disturbing symptoms of PTSD such as hypervigilance, anxiety, anger, and recurrent nightmares. If ketamine could be shown to be be a valuable treatment option for PTSD then this could have potentially large positive ramifications for the treatment of PTSD in America's veteran population.

Ketamine has historically been used as a dissociative anesthetic in emergency departments, operating rooms, and in austere military environments. It is a proven medication with a reassuring safety profile. This current study seeks to add to the body of knowledge regarding ketamine therapy by specifically looking at the combat veteran population. Eligible veterans will undergo the standard six-infusion Induction Series of ketamine infusions at Klarisana in San Antonio, Texas. Klarisana is a healthcare center which offers outpatient ketamine infusion therapy for the treatment of severe depression, PTSD, and various chronic pain conditions such as rheumatoid arthritis, fibromyalgia, neuropathy, and migraine headaches. Klarisana serves patients from all over south Texas including Austin, Houston, San Antonio, and Corpus Christi.

Patients who enroll in the current PTSD study will receive a standard battery of survey instruments which Klarisana implements before and after a series of infusions. These instruments will assess each patient's level of depression, degree of PTSD symptoms, as well as their use of alcohol and recreational drugs. The specific instruments are the...

Patient Health Questionnaire (PHQ-9) PTSD Checklist (PCL-5) Drug Abuse Screening Test (DAST-10) Alcohol Use Disorders Identification Test (AUDIT)

The investigator's goal is to formally analyze what changes may occur the participants' symptoms of PTSD and try to better establish the role which ketamine infusion therapy may play in the treatment of PTSD in the combat veteran population.

ELIGIBILITY:
Inclusion Criteria:

* The Veteran must be medically screened by Klarisana and be an appropriate candidate for ketamine therapy
* The Veteran must be between the ages of 18 and 75. The study is open to men and women.
* The Veteran must be able to speak and read the English language
* The Veteran must have a diagnosis of post-traumatic stress disorder assigned by the Department of Veterans Affairs. Veterans of a foreign military are also eligible but they must have been diagnosed with PTSD by the equivalent veteran healthcare organization in their country of military service
* The Veteran must have served in the US Military or a foreign military service in a designated combat zone. Documentation by a DD214 or equivalent is required
* The PTSD that The Veteran is suffering from has to have been caused by service in combat
* The PTSD that the Veteran is suffering from must be exerting a significant negative effect on his/her life

Exclusion Criteria:

* The Veteran must NOT be taking lamotrigine (Lamictal) or any monoamine oxidase inhibitor antidepressants
* The Veteran must not be currently enrolled in any other studies offering therapy for PTSD
* Veteran may NOT have uncontrolled blood pressure or congestive heart failure
* Veteran may NOT have a diagnosis of psychosis or any diagnosis on the psychosis spectrum

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans of the United States or foreign militaries who have served in combat and who now suffer from post traumatic stress disorder as a result of that military service.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Participant score on the PTSD Checklist - 5 (PCL-5) after a series of six ketamine infusions. | 3 weeks
  The PCL-5 is a twenty question survey instrument which is used to quantify the level of symptomatology in participants with post-traumatic stress disorder.

SECONDARY OUTCOMES:
Participant score on the Patient Health Questionnaire - 9 (PHQ-9) after a series of six ketamine infusions. | 3 weeks
  The PHQ-9 is a nine-question survey instrument which is used to quantify the level of depressive symptoms in participants.
Participant score on the Drug Abuse Screening Test (DAST-10) after a series of six ketamine infusions. | 3 weeks
  The DAST-10 is a ten-question self-report survey instrument which is used to assess participants' use of illicit drugs.
Participant score on the Alcohol Use Disorders Identification Test (AUDIT) after a series of six ketamine infusions. | 3 weeks
  The AUDIT is a ten-question self-reporting survey instrument which is used to identify participants' use of and potential dependence on alcohol

CONTACTS AND LOCATIONS:
Locations (1):
- Klarisana, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Murrough JW, Soleimani L, DeWilde KE, Collins KA, Lapidus KA, Iacoviello BM, Lener M, Kautz M, Kim J, Stern JB, Price RB, Perez AM, Brallier JW, Rodriguez GJ, Goodman WK, Iosifescu DV, Charney DS. Ketamine for rapid reduction of suicidal ideation: a randomized controlled trial. Psychol Med. 2015 Dec;45(16):3571-80. doi: 10.1017/S0033291715001506. Epub 2015 Aug 12. PMID 26266877
- [Background] McGowan JC, LaGamma CT, Lim SC, Tsitsiklis M, Neria Y, Brachman RA, Denny CA. Prophylactic Ketamine Attenuates Learned Fear. Neuropsychopharmacology. 2017 Jul;42(8):1577-1589. doi: 10.1038/npp.2017.19. Epub 2017 Jan 27. PMID 28128336
- [Background] Brachman RA, McGowan JC, Perusini JN, Lim SC, Pham TH, Faye C, Gardier AM, Mendez-David I, David DJ, Hen R, Denny CA. Ketamine as a Prophylactic Against Stress-Induced Depressive-like Behavior. Biol Psychiatry. 2016 May 1;79(9):776-786. doi: 10.1016/j.biopsych.2015.04.022. Epub 2015 May 4. PMID 26037911
- [Background] Burbiel JC. Primary prevention of posttraumatic stress disorder: drugs and implications. Mil Med Res. 2015 Oct 26;2:24. doi: 10.1186/s40779-015-0053-2. eCollection 2015. PMID 26504586
- [Background] Fortea A, Espinosa L, Oliveras C, Bruguera P, Benabarre A. Ketamine associated with electroconvulsive therapy for treatment-resistant depression in the elderly: Two case reports. Rev Psiquiatr Salud Ment. 2017 Apr-Jun;10(2):125-126. doi: 10.1016/j.rpsm.2016.12.001. Epub 2017 Feb 10. No abstract available. English, Spanish. PMID 28209259
- [Background] Witkin JM, Mitchell SN, Wafford KA, Carter G, Gilmour G, Li J, Eastwood BJ, Overshiner C, Li X, Rorick-Kehn L, Rasmussen K, Anderson WH, Nikolayev A, Tolstikov VV, Kuo MS, Catlow JT, Li R, Smith SC, Mitch CH, Ornstein PL, Swanson S, Monn JA. Comparative Effects of LY3020371, a Potent and Selective Metabotropic Glutamate (mGlu) 2/3 Receptor Antagonist, and Ketamine, a Noncompetitive N-Methyl-d-Aspartate Receptor Antagonist in Rodents: Evidence Supporting the Use of mGlu2/3 Antagonists, for the Treatment of Depression. J Pharmacol Exp Ther. 2017 Apr;361(1):68-86. doi: 10.1124/jpet.116.238121. Epub 2017 Jan 30. PMID 28138040
- [Background] Murrough JW, Burdick KE, Levitch CF, Perez AM, Brallier JW, Chang LC, Foulkes A, Charney DS, Mathew SJ, Iosifescu DV. Neurocognitive effects of ketamine and association with antidepressant response in individuals with treatment-resistant depression: a randomized controlled trial. Neuropsychopharmacology. 2015 Mar 13;40(5):1084-90. doi: 10.1038/npp.2014.298. PMID 25374095
- See also: For more information on the study sponsor - Klarisana — http://klarisana.com